CLINICAL TRIAL: NCT05077007
Title: Evaluation of Renal Damage After PCNL and ESWL Using Novel RNA Based Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Science,Technology & Innovation Funding Authority (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FMASU R 77/ 2021
Record Dates: First submitted 2021-08-31; First posted 2021-10-13 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-04

CONDITIONS: Acute Kidney Injury; Renal Calculi; Percutaneous Nephrolithotomy; Extracorporeal Shockwave Lithotripsy
Keywords: lncRNA, mRNA, ESWL,PCNL,SBF2-AS1, FENDRR-19, NLRP3.
MeSH Terms: conditions — Acute Kidney Injury; Kidney Calculi | interventions — Nephrolithotomy, Percutaneous; Lithotripsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Percutaneous nephrolithotomy (Active Comparator): patients suffering of pelvic renal stones underwent Percutaneous nephrolithotomy
  Interventions: Procedure: Percutaneous nephrolithotomy
- Extracorporeal Shock Wave Lithotripsy (Active Comparator): patients suffering of pelvic renal stones underwent Extracorporeal Shock Wave Lithotripsy
  Interventions: Procedure: Extracorporeal Shock Wave Lithotripsy
- control group (No Intervention): Healthy volunteers with negative history of renal stones or renal impairment to measure the level of urinary markers in their urine samples

INTERVENTIONS:
Procedure: Percutaneous nephrolithotomy — Endoscopic stone Extraction from the kidney by making a puncture and dilate a tract direct into the kidney through muscle wall and renal parenchyma
  Other Names: PCNL
  Arms: Percutaneous nephrolithotomy
Procedure: Extracorporeal Shock Wave Lithotripsy — Using Shock waves from outside the body targeted at a kidney stone causing the stone to fragment. The stones are broken into tiny pieces.
  Other Names: ESWL
  Arms: Extracorporeal Shock Wave Lithotripsy

SUMMARY:
The study evaluate the damage effect of ESWL and PCNL on kidney tissue by measuring non-coding lnc-RNA profile in urine before and after ESWL and PCNL procedures

DETAILED DESCRIPTION:
The study evaluate the damage effect of ESWL and PCNL on kidney tissue by measuring non-coding lnc-RNA profile in urine before and after ESWL and PCNL procedures and assess their usefulness as diagnostic biomarkers for AKI and the relationship between the selected RNA based biomarker panel and clinicopathological changes of patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients :

  1. Patients undergoing treatment for a stone(s) located in the kidney less than 2 cm
  2. Radiopaque stone
  3. Able and willing to give informed consent

Inclusion criteria for Healthy volunteers

1. No history of kidney or stone disease
2. Asymptomatic
3. No indwelling ureteral stent
4. Willing to provide medical history information
5. Able and willing to give informed consent

Exclusion Criteria:

* Exclusion criteria for patients

  1. Active urinary tract infection
  2. Bleeding disorder
  3. Chronic renal failure (eGFR<30)
  4. Ureteral stone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-22 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of renal damage after PCNL and ESWL using novel RNA based Biomarkers | Before the procedure by 2hours and after the procedure by 2 and 24 hours
  Evaluation of kidney injury after procedures PCNL and ESWL by measuring the change of the level of novel non-coding lnc-RNA profile in urine

CONTACTS AND LOCATIONS:
Overall Officials: waleed Mousa, Principal Investigator — Urology Department, Ain Shams University, Abassia, Cairo
Locations (1):
- Urology Department, Faculty of Medicine, Ain Shams University, Cairo, Egypt